CLINICAL TRIAL: NCT02712853
Title: Improving Autism Screening With Brain-Related miRNA
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Steven Hicks, Assistant Professor of Pediatrics, Milton S. Hershey Medical Center
Other Study IDs: Study00003658
Record Dates: First submitted 2016-02-08; First posted 2016-03-18 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Autism Spectrum Disorder; Developmental Delay
MeSH Terms: conditions — Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Salivary RNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Autism Spectrum Disorder (ASD): Age at enrollment: 18 months to 6 years with established DSM-5 diagnosis of autism spectrum disorder. Exclusion criteria include:
  wards of the state syndromic autism (attributed to a known genetic mutation) active periodontal infection active upper respiratory infection
  Interventions: Other: Saliva collection; Other: Vineland Adaptive Behavior Scale-II Assessment
- Control: Age 18 months to 6 years without autism spectrum disorder (may have typical development or developmental delay without autism - as defined by negative MCHAT-R or negative ADOS-II evaluation)
  Exclusion criteria include:
  wards of the state active periodontal infection active upper respiratory infection
  Interventions: Other: Saliva collection; Other: Vineland Adaptive Behavior Scale-II Assessment

INTERVENTIONS:
Other: Saliva collection — Collection of saliva via swab for miRNA processing
Other: Vineland Adaptive Behavior Scale-II Assessment

SUMMARY:
The goal of this project is to identify specific miRNAs that are increased or decreased in the saliva of children with developmental delay and are useful for screening toddlers for ASD. Such a screening tool would improve the specificity of diagnosis, streamline referrals to developmental specialists, and expedite the arrangement of early intervention services.

DETAILED DESCRIPTION:
The central aim of this project is to characterize the expression of exosomal microRNA (miRNA) in children with autism spectrum disorder (ASD). Currently, the CDC estimates the prevalence of ASD in U.S. children to be 1 in 68. Yet, the biological causes, diagnosis, and treatment of this disease remain ambiguous. Growing evidence implicates a genetic role in ASD. miRNAs regulate genetic expression and are altered in lymphocytes, neurons and serum of patients with ASD. Recent studies of miRNAs have shown that they can be packaged into exosomal vessels and extruded from neurons as extracellular signaling tools. This knowledge provides a novel approach for examining the genetic regulation of the central nervous system.

We propose to measure the expression of extracellular miRNA in children with ASD. Expression levels of miRNA from blood and saliva will be compared between children with autism and normally developing controls. The goal of this study will be to identify genetic regulatory mechanisms involved in ASD and provide potential biomarkers for diagnostic screening.

The primary endpoints of this study are as follows:

1. Characterization of brain-related miRNA in the saliva of children with ASD and typically developing control children between the ages of two and five years.
2. Identification of sets of miRNAs in saliva and plasma that are predictive of both ASD diagnosis and severity of ASD symptoms. This aim will enroll ASD and control children age 12-24 months (inclusive).

Secondary endpoints include the identification of miRNA expression patterns that correlate with ASD symptom severity measured with standardized neuropsychologic testing and to characterize parental knowledge and attitudes towards epigenetic testing in the context of ASD..

ELIGIBILITY:
Inclusion Criteria:

* • Age at enrollment: 18 months and 6 years (inclusive)

  * Control group documented negative ASD screening on M-CHAT-R
  * ASD group: established DSM-5 diagnosis
  * Parent/guardian must be fluent in written and spoken English (required to complete study specific questionnaires etc)

Exclusion Criteria:

For autistic subjects study exclusion criteria will include:

• Autistic subjects with known syndromic autism (attributed to a known genetic mutation)

Control subjects only exclusion criteria will include:

• A diagnosis of autism

For both groups: wards of the state, active periodontal infection, active upper respiratory infection

Ages: 18 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will compare salivary miRNA in 2 groups of children between the ages of 18 months and 6 years, 11 months of age:
  Group 1: Children with autism spectrum disorder (ASD), diagnosed by a qualified clinical specialist using DSM-5 criteria and confirmed with ADOS, CASD, or some additional semi-structured evaluation measure. ASD will not be attributable to an underlying genetic phenotype.
  Group 2: Healthy controls with negative MCHAT-R screening not meeting DSM-5 criteria for ASD
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
salivary miRNA profile | at time of collection (between 18 months and 6 years of age)
  Measures of miRNA abundance in saliva

SECONDARY OUTCOMES:
Measures of adaptive function | at time of enrollment (between 18 months and 6 years)
  Vineland adaptive behavior composite score
Measure of autistic behavior | at time of enrollment (between 18 months and 6 years)
  Autism Diagnostic Observation Schedule (ADOS) Composite Score (when clinically indicated)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hicks, MD, PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available

REFERENCES:
- [Background] Mundalil Vasu M, Anitha A, Thanseem I, Suzuki K, Yamada K, Takahashi T, Wakuda T, Iwata K, Tsujii M, Sugiyama T, Mori N. Serum microRNA profiles in children with autism. Mol Autism. 2014 Jul 30;5:40. doi: 10.1186/2040-2392-5-40. eCollection 2014. PMID 25126405
- [Background] Sarachana T, Zhou R, Chen G, Manji HK, Hu VW. Investigation of post-transcriptional gene regulatory networks associated with autism spectrum disorders by microRNA expression profiling of lymphoblastoid cell lines. Genome Med. 2010 Apr 7;2(4):23. doi: 10.1186/gm144. PMID 20374639
- [Background] Abu-Elneel K, Liu T, Gazzaniga FS, Nishimura Y, Wall DP, Geschwind DH, Lao K, Kosik KS. Heterogeneous dysregulation of microRNAs across the autism spectrum. Neurogenetics. 2008 Jul;9(3):153-61. doi: 10.1007/s10048-008-0133-5. Epub 2008 Jun 19. PMID 18563458